CLINICAL TRIAL: NCT05339711
Title: Investigation of Physiological and Psychological Effects of Robotic Cat and Betta Fish Therapies in Hemodialysis Patients: A Randomized Controlled Study
Brief Title: Effects of Robotic Cat and Betta Fish Therapies in Hemodialysis Patients
Acronym: Pet Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Lecturer, Ph.D, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCS09042022
Record Dates: First submitted 2022-04-09; First posted 2022-04-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hemodialysis; Animal Assisted Therapy; Adaptation; Happiness; Loneliness; Symptom
Keywords: Adaptation; Happiness; Hemodialysis; Loneliness; Pet therapy; Symptom
MeSH Terms: interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Power analysis was performed in the selection of patients to be sampled. The number of samples, the G*Power program 3.1.9.6 error rate α=0.05, and due to the lack of work he has done on the subject before in different populations (old) (32) pet therapy is a targeted domain 0.475 three groups (robot kedi grubu, Betta balık grubu, kontrol grubu) by reference to the size and power of test work is 0.80 (80%), while for a group of three in total, 48 (16 for each group) patients was calculated. Considering situations such as wanting to leave the study or death during the study, each group was increased by 10% and a total of 54 patients were included in the study, 18 patients for each group.
Masking Description: While the patients were randomized; In order to keep the possibility of being affected by each other at a minimum level, the study was continued with the same application group in the same session group. For example; It's like working only with the robot cat group in the 08:00-12:00 session group on Mondays. In order to reduce the possibility of selection bias due to sample selection, "single-stage cluster type random sampling", which is a subtype of random sampling, was used. In addition, before the study, patients were informed about the study and their consent was obtained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robotic Pet Therapy/Robot Cat Group (Experimental): In the robot cat group, the patients were given face-to-face personal information about the robot cat for about 15 minutes in the waiting room by the researcher, and the "Robot Cat Information Brochure" was given. Therefore, in this study, the patients interacted with the robot cat "Silver" for 20 minutes during the hemodialysis session once a week for eight weeks (two months) under the supervision of the researcher. After eight weeks of robotic pet therapy in the hemodialysis unit, this group of patients was followed up by the researcher with the same applications, without robotic pet therapy for eight more weeks. Data collection tools were applied to this group of patients before the study. Again, in the last week of the 1st, 2nd, 3rd and 4th months of the study, all other data collection tools were applied, except the "Structured Patient Information Form".
  Interventions: Other: Robotic Pet Therapy/Robot Cat Group
- Pet Therapy/Betta Fish Group (Experimental): In the Betta fish group, the patients were given a 15-minute hands-on, face-to-face, individual information about Betta fish care in the waiting room by the researcher, and a "Betta Fish Information Brochure" was given to the patients. Then, the patients were asked to take care of the fish given to them at home for two months.This group of patients was given pet therapy for eight weeks, and then followed by the researcher with the same practices for another eight weeks without pet therapy. In order to observe or measure the positive effects of fish on patients, patients should spend at least 10 minutes with fish during the day (52). Data collection tools were applied to this group of patients before the study. Again, in the last week of the 1st, 2nd, 3rd and 4th months of the study, all other data collection tools were applied, except the "Structured Patient Information Form".
  Interventions: Other: Pet Therapy/Betta Fish Group
- Control Group (No Intervention): This group of patients was only informed about the study and received routine hemodialysis treatment. The patients were followed for four months. Data collection tools were applied to the patients before the study. Again, in the last week of the 1st, 2nd, 3rd and 4th months of the study, all other data collection tools were applied, except the "Structured Patient Information Form".

INTERVENTIONS:
Other: Robotic Pet Therapy/Robot Cat Group — İn this study, the patients interacted with the robot cat "Silver" for 20 minutes during the hemodialysis session once a week for eight weeks (two months) under the supervision of the researcher.
  Arms: Robotic Pet Therapy/Robot Cat Group
Other: Pet Therapy/Betta Fish Group — İn this study, two fish and the necessary materials (aquarium, fish food, plastic plant, aquarium stone, etc.) were given to the patients by the researcher to keep pets for eight weeks.
  Arms: Pet Therapy/Betta Fish Group

SUMMARY:
The research was carried out as a randomized controlled trial to examine the physiological and psychological effects of robotic cat and Betta fish therapies in hemodialysis patients.

DETAILED DESCRIPTION:
Along with the benefit of hemodialysis treatment, patients develop physical and psychosocial problems and symptoms associated with hemodialysis. Undesirable symptoms experienced by patients undergoing hemodialysis include hypotension/hypertension, respiratory distress, headache, back-chest pain, muscle cramps, nausea-vomiting, fatigue, fever, constipation, diarrhea, itching. In addition to negative feelings such as anger, anxiety, unhappiness and fear associated with hemodialysis, patients often experience adjustment disorder, anxiety, depression and sleep disorders, and may experience social isolation and loneliness with the fear of being a burden to their friends or family members. The physical symptoms that patients receiving hemodialysis treatment have to cope with and psychological symptoms such as unhappiness and loneliness make it difficult to adapt to their disease and contribute to an increase in mortality.

Today, "pet therapy" is used for treatment in many hospitals, psychiatry clinics, nursing homes and rehabilitation centers. Pet therapy is an application in the Nursing Interventions Classification. In studies with different animals on different populations in health services, hospitals, psychiatry clinics, nursing homes and rehabilitation centers, pet therapy; It is stated that it has physiological and psychological benefits such as decrease in psychiatric signs and symptoms, increase in cardiovascular system functionality, increase in socialization skills and individual self-management. It is reported that the physiological and psychological benefits of pet therapy applications have been proven in many of the studies using many animals (such as birds, dogs, cats, fish) and robot simulations. It has been reported that robotic pet therapy reduces depression, agitated behaviors, pain, stress hormone levels and loneliness, increases heart rate, happiness, and quality of life. Again, it is stated that even a simple movement of live animals reduces loneliness, anxiety, depression and social isolation in humans.

It has been determined that an unpublished experimental doctoral thesis study, of which a poster statement can be reached, was conducted abroad on the effect of "the effect of pet therapy with live dogs on depression" in patients with CRF. Again, one pilot study and one pre-test-post-test study were found in which the effect of pet therapy on happiness with a live dog was examined. In Turkey, no study was found with pet therapy in patients undergoing CRF and hemodialysis. However, there is limited information in the literature about the benefits of human-fish interactions related to pet therapy. It has been reported that ornamental betta fish increase individual self-management, and reduce anxiety and stress. In a systematic review, it was reported that various fish species reduced anxiety, physiological stress, anxiety and pain, provided relaxation, improved food intake, had positive benefits on mood and body weight (weight gain), but no information was found about loneliness.

About the subject, only pet therapy with live dogs was used in hemodialysis patients, and no experimental study was found. In addition, it was determined that there was no information about the effect of Betta fish therapy on loneliness and that happiness, dialysis symptoms, compliance with ESRD, and body mass index (BMI) were not examined before in patients undergoing hemodialysis. The fact that the mentioned parameters were not examined indicates that there is a lack of evaluation of robotic cat or Betta fish therapies. In line with this information, the aim of this study was to examine the positive physiological (dialysis symptoms, BMI) and psychological (dialysis symptoms, happiness, loneliness, adaptation to ESRD) effects of robotic cat and Betta fish therapies in patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 years old,
* Accepting to participate in the research,
* Being literate,
* Being able to communicate verbally,
* Receiving outpatient hemodialysis treatment three times a week in the same institution,
* Absence of any impairment in mental and cognitive functions,
* Weight and height measurements can be made while standing,
* Being on hemodialysis treatment for at least three months (33),
* Being able to perform self-care activities independently,
* Not having allergies for patients in the robot cat group,
* Desiring to spend time with the robotic cat "Silver" during hemodialysis by the patients in the robot cat group,
* Wanting to nutrition and care fish at home by patients in the betta fish group.

Exclusion Criteria:

* Refusal to participate in the research,
* Being on peritoneal dialysis,
* Being diagnosed with a psychiatric disorder diagnosed by a psychiatrist,
* Unstable general condition (hemodynamically) (heart rate <60 beats/min, systolic blood pressure <100 mm/Hg or diastolic blood pressure <60 mm/Hg),
* Patients with chronic obstructive pulmonary disease (COPD) (except Mild COPD Stage 1) and advanced heart failure were identified (34, 35).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Body mass İndex Monitoring | 16 week
  This form includes BMI, an anthropometric measurement. To obtain the Body Mass Index, the patient's body weight (kg) was divided by the square of the height (m) (BMI=kg/m2).
  Before the research, 5 measurements were made, twice in the 1st month and 2nd month when pet therapy was applied, and twice in the two-month follow-up after the pet therapy application was terminated.
De Jong Gierveld Loneliness Scale | 16 week
  The scale was first developed by De Jong Gierveld and Kamphuis in 1985. The Turkish adaptation of the scale with factor loadings between 0.64-0.86 was carried out by Çavdar, Bağcı, Chorbaci, Saritas and Tasdelen in 2015. Social loneliness and emotional loneliness two sub-scale in size 11 items in Scale. It is a four-point likert (4=Very convenient, 3=Convenient, 2=Not convenient, 1=Not convenient at all) type scale. Since the items in the social loneliness dimension contain positive statements, these items are reverse items. As the score obtained from the scale increases, the levels of loneliness increase.
  Before the research, 5 measurements were made, twice in the 1st month and 2nd month when pet therapy was applied, and twice in the two-month follow-up after the pet therapy application was terminated.
Subjective Happiness Scale (SHS) | 16 week
  Developed by Lyubomirsky and Lepper, SHD is a seven-point Likert type, self-report style. The scale consists of four items; Since the fourth item contains a negative statement, this item is the reverse item. The lowest score taken from the scale is four, the highest score is 28, and as the individual's scale score increases, the level of happiness increases.
  Before the research, 5 measurements were made, twice in the 1st month and 2nd month when pet therapy was applied, and twice in the two-month follow-up after the pet therapy application was terminated.
End Stage Renal Disease (ESRD)-Adherence Questionnaire | 16 week
  This scale was developed by Kim, Evangelista, Phillips, Pavlish, and Kopple. The ESRD-Adaptation Scale consists of four compliance behaviors subscales: participation in treatment (1st, 3rd and 5th items), medicine use (6th item), fluid restriction (8th item), and dietary restriction (9th item). Items 2, 5 and 7 of the items do not have a point value. The range of scores that can be obtained from the scale is between 0-1200, and as the score increases, the compliance of the patients with the treatment also increases.
  Before the research, 5 measurements were made, twice in the 1st month and 2nd month when pet therapy was applied, and twice in the two-month follow-up after the pet therapy application was terminated.
Dialysis Symptom Index (DSİ) | 16 week
  Weisbord et al. has a total of 30 items in which both emotional and physical symptoms of dialysis patients and the severity of these symptoms are evaluated. After the patients answered yes-no to the questions regarding the symptoms they experienced within a week, their symptoms with a yes answer are re-evaluated in a five-point Likert type ("5 points: A lot", "4 points: Very little", "3 points: Sometimes", "2 points: A little", "1 point: Not at all"). The total score to be obtained from the scale ranges from 0 to 150.
  Before the research, 5 measurements were made, twice in the 1st month and 2nd month when pet therapy was applied, and twice in the two-month follow-up after the pet therapy application was terminated.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Tecnical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll decide later

REFERENCES:
- [Derived] Demirag H, Hintistan S. Investigation of physiological and psychological effects of robotic cat and betta fish therapies in hemodialysis patients: A randomized controlled study. Complement Ther Clin Pract. 2022 Nov;49:101647. doi: 10.1016/j.ctcp.2022.101647. Epub 2022 Jul 31. PMID 35932699